CLINICAL TRIAL: NCT03341156
Title: Optimized Administration of Prothrombin Complex Concentrate (PCC) vs. Standard Transfusion During/After Heart Transplantation - OPSTAHT
Brief Title: Administration of Prothrombin Complex Concentrate vs. Standard Transfusion During/After Heart Transplantation
Acronym: OPSTAHT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Standard practice change prohibited enrollment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020099
Record Dates: First submitted 2017-08-28; First posted 2017-11-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Heart Disease End Stage; Heart Failure，Congestive
Keywords: Heart transplantation
MeSH Terms: conditions — Heart Failure | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Kcentra (PCC) (Experimental): Half of subjects enrolled will be randomized to the Kcentra (PCC) group.
  Interventions: Drug: Kcentra
- Frozen Plasma Product, Human (Active Comparator): Half of subjects enrolled will be randomized to the standard transfusion group and receive fresh frozen plasma intra-operatively.
  Interventions: Drug: Frozen Plasma Product, Human

INTERVENTIONS:
Drug: Kcentra — Kcentra will be administered in 2 divided doses; Pre-bypass (5-10 units/kg based on body weight and preoperative INR and post-protamine based of the pre-bypass dose and the preoperative INR; daily maximum dose not to exceed 5000 IU (50 IU/kg)
  Other Names: prothrombin complex concentrate
  Arms: Kcentra (PCC)
Drug: Frozen Plasma Product, Human — If the patient is randomized to receive standard transfusion they will receive 2 U of fresh frozen plasma intravenously before cardiopulmonary bypass and then up to 4-8 U of plasma added to the cardiopulmonary bypass reservoir during rewarming.
  Other Names: Fresh Frozen Plasma
  Arms: Frozen Plasma Product, Human

SUMMARY:
This study is comparing the use of Kcentra vs. standard transfusion in patients undergoing heart transplantation surgery. Half of the patients will receive Kcentra, while the other half will receive fresh frozen plasma.

DETAILED DESCRIPTION:
This study will be a randomized (1:1; PCC vs. plasma), open-label trial of hemostatic therapies during heart transplantation. The goal is to enroll 60 patients. Informed consent will be obtained from patients meeting the inclusion and exclusion criteria before the initiation of any study specific procedures. Eligible patients will be randomized to receive either PCC or plasma transfusion. The efficacy of interventions will be evaluated after 30 minutes of protamine administration. After the heart transplantation, thrombocytopenia and/or hypofibrinogenemia may worsen bleeding associated with vitamin K dependent factor deficiencies. Transfusion of platelets and/or cryoprecipitate is permitted if abnormal laboratory values are observed during the rewarming phase of CPB; platelet count <100 x 103/µl, and fibrinogen <200 mg/dl, respectively. Laboratory tests (hematocrit, platelet count, PT, PTT, POC-PT, coagulation factor and inhibitor levels (e.g., factor II, antithrombin), thromboelastometry or thromboelastography, endogenous thrombin generation) will also be obtained at baseline, twice during surgery and at 12-24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent.
* Be at least 18 years of age.
* Patients with or without ventricular assist device (VAD) undergoing heart transplantation
* Patients who have been on warfarin for at least 72 hours before cardiopulmonary bypass procedures for heart transplantation.
* International normalization ration (INR) greater than or equal to 1.5
* Body temperature greater than 35.0 degrees Celsius.
* Blood pH greater than 7.2
* Hemoglobin greater than 7.0 mg/dL.

Exclusion Criteria:

* Treatment with clopidogrel, prasugrel, or ticagrelor within 5 days prior to study surgery.
* Known or suspected thrombophilia such as factor V Leiden, hereditary antithrombin III deficiency, heparin-induced thrombocytopenia, disseminated intravascular coagulation.
* Ischemic or thromboembolic events within 6 weeks of study surgery.
* Known allergy/anaphylaxis to prothrombin complex concentrate or albumin.
* Any indication that a potential subject did not comprehend the study restrictions, procedures. or consequences therein an informed consent cannot be convincingly given.
* Patients on respiratory support including extracorporeal membrane oxygenation (ECMO) .
* Life expectancy less than 48 hours.
* Excluded at the discretion of the surgeon based upon surgical safety precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Amount of Chest Tube Drainage | From patient out of room time until 24 hours after
  Primary outcome: Amount of chest tube output in the first 24 hours

SECONDARY OUTCOMES:
Postoperative INR | 30 Minutes post-treatment (after the last dose is completed)
  INR value
Blood Product Use | In OR (from OR entry to OR out of room time); postoperatively (patient out of room time) to 24 hours after; from 24 hours after until 30 days post surgery or until discharge (whichever comes first)
  Total hemostatic blood product use including plasma, platelets, cryoprecipitate, and recombinant activated factor VII.
Red Blood Cell Use | Intraoperatively(from start of first intervention until start of second intervention;after 2nd intervention(post-bypass)until patient out of room time) & Postoperatively(from patient out of room time until 24 hours after;24 hours after until 30 days)
  Red Blood Cell Use Intraoperatively and Postoperatively
Need for circulatory support | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who needed circulatory support (ECMO or VAD)
Mechanical Ventilation | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who needed mechanical ventilation for more than 72 hours
Tracheostomy | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who needed a tracheostomy
Renal Failure | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who experience renal failure requiring dialysis
Sepsis | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who experienced sepsis infection morbidity consisted of sepsis syndrome, septic shock, or mediastinitis. In addition, the diagnosis of sepsis included organisms isolated from the cultures along with elevated temperature and white blood cell counts.
Death | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who died
Stroke or postoperative neurological dysfunction | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who experienced a stroke or postoperative neurological dysfunction (seizures, delirium, unconsciousness, encephalopathy)
Gastrointestinal complication requiring bowel resection | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who experienced gastrointestinal complications requiring bowel resection
Peripheral vascular complication | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who experience peripheral vascular complications requiring surgery (thrombectomy, bypass, and amputations)
Deep Vein Thrombosis and Pulmonary Thromboembolism | 30 days post-operative or until discharge (whichever comes first)
  Percentage of patients who develop a deep vein thrombosis and/ or pulmonary thromboembolism
Plasma Coagulation Factor levels | At baseline, post-bypass/pre-protamine, 30 minutes post-protamine, 12-24 hours post treatment
  Plasma coagulator factor levels will be analyzed via blood laboratory tests
Thrombin Generation Assay | At baseline, post-bypass/pre-protamine, 30 minutes post-protamine, 12-24 hours post treatment
  Thrombin Generation assay will be analyzed via blood laboratory tests
Surgical Re-exploration | 30 days post-operative or until discharge (whichever comes first)
  Surgical Re-Exploration that is related to heart transplant surgery

OTHER OUTCOMES:
Direct Cost Benefit | From infusion until 30 days post heart transplant
  Acquisition costs for test agents and blood bank related charges (thawing, etc.)
Total surgical time | From anesthesia start time until anesthesia stop time
  Total time of surgical duration will be measured in the corresponding time frame
Time to hospital discharge | From patient out of room time to hospital discharge (or 30 days post heart transplant, whichever comes first)
  Time until discharge from the hospital post study intervention will be measured
Time to Intensive Care Unit (ICU) discharge | From patient out of room time to ICU discharge (or 30 days post heart transplant, whichever comes first)
  Time until discharge from the ICU post study intervention will be measured
Indirect Cost Benefits | From last intervention/infusion until 30 days post heart transplant or until discharge
  Extra costs related to study drug (PCC and plasma) related complications (volume overload, thrombotic complications)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Tanaka, MD, Principal Investigator — University of Maryland, Baltimore; Kathirvel Surbramaniam, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - Upmc Presbyterian Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolliger D, Gorlinger K, Tanaka KA. Pathophysiology and treatment of coagulopathy in massive hemorrhage and hemodilution. Anesthesiology. 2010 Nov;113(5):1205-19. doi: 10.1097/ALN.0b013e3181f22b5a. PMID 20881594
- [Background] Mathias T, Puca KE, Downey F, Boyle AJ: Use of Vitamin K and Prothrombin Complex Concentrate as Warfarin Reversal Prior to Heart Transplant. Journal of Heart and Lung Transplantation 2012; 31: S154
- [Background] Kantorovich A, Fink JM, Militello MA, Wanek MR, Smedira NG, Soltesz EG, Moazami N. Low-dose 3-factor prothrombin complex concentrate for warfarin reversal prior to heart transplant. Ann Pharmacother. 2015 Aug;49(8):876-82. doi: 10.1177/1060028015585344. Epub 2015 May 18. PMID 25986007
- [Background] Marshall AL, Levine M, Howell ML, Chang Y, Riklin E, Parry BA, Callahan RT, Okechukwu I, Ayres AM, Nahed BV, Goldstein JN. Dose-associated pulmonary complication rates after fresh frozen plasma administration for warfarin reversal. J Thromb Haemost. 2016 Feb;14(2):324-30. doi: 10.1111/jth.13212. Epub 2016 Feb 2. PMID 26644327
- [Background] Demeyere R, Gillardin S, Arnout J, Strengers PF. Comparison of fresh frozen plasma and prothrombin complex concentrate for the reversal of oral anticoagulants in patients undergoing cardiopulmonary bypass surgery: a randomized study. Vox Sang. 2010 Oct;99(3):251-60. doi: 10.1111/j.1423-0410.2010.01339.x. PMID 20840339
- [Background] Tanaka KA, Mazzeffi MA, Grube M, Ogawa S, Chen EP. Three-factor prothrombin complex concentrate and hemostasis after high-risk cardiovascular surgery. Transfusion. 2013 Apr;53(4):920-1. doi: 10.1111/trf.12110. No abstract available. PMID 23565996
- [Background] Song HK, Tibayan FA, Kahl EA, Sera VA, Slater MS, Deloughery TG, Scanlan MM. Safety and efficacy of prothrombin complex concentrates for the treatment of coagulopathy after cardiac surgery. J Thorac Cardiovasc Surg. 2014 Mar;147(3):1036-40. doi: 10.1016/j.jtcvs.2013.11.020. Epub 2013 Dec 22. PMID 24365268
- [Background] Rao VK, Lobato RL, Bartlett B, Klanjac M, Mora-Mangano CT, Soran PD, Oakes DA, Hill CC, van der Starre PJ. Factor VIII inhibitor bypass activity and recombinant activated factor VII in cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1221-6. doi: 10.1053/j.jvca.2014.04.015. PMID 25281040
- [Background] Balsam LB, Timek TA, Pelletier MP. Factor eight inhibitor bypassing activity (FEIBA) for refractory bleeding in cardiac surgery: review of clinical outcomes. J Card Surg. 2008 Nov-Dec;23(6):614-21. doi: 10.1111/j.1540-8191.2008.00686.x. Epub 2008 Sep 10. PMID 18793226
- [Background] Ortmann E, Besser MW, Sharples LD, Gerrard C, Berman M, Jenkins DP, Klein AA. An exploratory cohort study comparing prothrombin complex concentrate and fresh frozen plasma for the treatment of coagulopathy after complex cardiac surgery. Anesth Analg. 2015 Jul;121(1):26-33. doi: 10.1213/ANE.0000000000000689. PMID 25822921
- [Background] Goldstein JN, Refaai MA, Milling TJ Jr, Lewis B, Goldberg-Alberts R, Hug BA, Sarode R. Four-factor prothrombin complex concentrate versus plasma for rapid vitamin K antagonist reversal in patients needing urgent surgical or invasive interventions: a phase 3b, open-label, non-inferiority, randomised trial. Lancet. 2015 May 23;385(9982):2077-87. doi: 10.1016/S0140-6736(14)61685-8. Epub 2015 Feb 27. PMID 25728933
- [Background] Tanaka KA, Mazzeffi MA, Strauss ER, Szlam F, Guzzetta NA. Computational simulation and comparison of prothrombin complex concentrate dosing schemes for warfarin reversal in cardiac surgery. J Anesth. 2016 Jun;30(3):369-76. doi: 10.1007/s00540-015-2128-3. Epub 2016 Jan 9. PMID 26749482
- [Background] Sarode R, Milling TJ Jr, Refaai MA, Mangione A, Schneider A, Durn BL, Goldstein JN. Efficacy and safety of a 4-factor prothrombin complex concentrate in patients on vitamin K antagonists presenting with major bleeding: a randomized, plasma-controlled, phase IIIb study. Circulation. 2013 Sep 10;128(11):1234-43. doi: 10.1161/CIRCULATIONAHA.113.002283. Epub 2013 Aug 9. PMID 23935011
- [Background] Subramaniam K. Early graft failure after heart transplantation: prevention and treatment. Int Anesthesiol Clin. 2012 Summer;50(3):202-27. doi: 10.1097/AIA.0b013e3182603ead. No abstract available. PMID 22735727
- [Background] Tholpady A, Monson J, Radovancevic R, Klein K, Bracey A. Analysis of prolonged storage on coagulation Factor (F)V, FVII, and FVIII in thawed plasma: is it time to extend the expiration date beyond 5 days? Transfusion. 2013 Mar;53(3):645-50. doi: 10.1111/j.1537-2995.2012.03786.x. Epub 2012 Jul 15. PMID 22803679
- [Background] Scott E, Puca K, Heraly J, Gottschall J, Friedman K. Evaluation and comparison of coagulation factor activity in fresh-frozen plasma and 24-hour plasma at thaw and after 120 hours of 1 to 6 degrees C storage. Transfusion. 2009 Aug;49(8):1584-91. doi: 10.1111/j.1537-2995.2009.02198.x. PMID 19413730
- [Background] Karkouti K, McCluskey SA, Syed S, Pazaratz C, Poonawala H, Crowther MA. The influence of perioperative coagulation status on postoperative blood loss in complex cardiac surgery: a prospective observational study. Anesth Analg. 2010 Jun 1;110(6):1533-40. doi: 10.1213/ANE.0b013e3181db7991. Epub 2010 Apr 30. PMID 20435945